CLINICAL TRIAL: NCT01657409
Title: Comparison of the Therapeutic Effects of Different Injection Number of the Same Dose of Botulinum Toxin A on Overactive Bladder Syndrome
Brief Title: Different Injection Number of the Same Dose of Botulinum Toxin A on Overactive Bladder Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Department of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCGHUROL003
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Overactive Bladder
Keywords: botulinum toxin; detrusor overactivity
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Patients were randomized to receive different injection number of onabotulinumtoxinA
Who Masked: Participant
Masking Description: Participants did not aware how many injections were performed
Oversight: Data Monitoring Committee: No

ARMS (3):
- BoNT-A (10 injection) (Experimental): 100 U in 10ml, 1.0ml for each injection, totally 10 injections at bladder body
  Interventions: Drug: BoNT-A (10 injection)
- BoNT-A (20 injections) (Experimental): 100 U in 10ml, 0.5ml for each injection, totally 20 injections at bladder body
  Interventions: Drug: BoNT-A (20 injection)
- BoNT-A (40 injections) (Experimental): 100 U in 10ml, 0.25ml for each injection, totally 40 injections at bladder body
  Interventions: Drug: BoNT-A (40 injection)

INTERVENTIONS:
Drug: BoNT-A (10 injection) — BoNT-A 100 U 10 injections
  Other Names: Botulinum Toxin A (Botox)
  Arms: BoNT-A (10 injection)
Drug: BoNT-A (20 injection) — BoNT-A 100 U 20 injections
  Other Names: Botulinum Toxin A (Botox)
  Arms: BoNT-A (20 injections)
Drug: BoNT-A (40 injection) — BoNT-A 100 U 40 injections
  Other Names: Botulinum Toxin A (Botox)
  Arms: BoNT-A (40 injections)

SUMMARY:
Overactive bladder (OAB) is a symptom syndrome characterized by urgency frequency with or without urge urinary incontinence (UUI) that may affect the patients' quality of life. Current medical treatments are usually unsuccessful in completely eradicating urgency sensation. Intra-detrusor injection of botulinum toxin A (BoNT-A) modulates the release of neurotransmitters from sensory nerve endings and effectively modulates the inflammatory process mediated by nociceptive afferent nerve dysfunction. Satisfactory clinical results were achieved with intravesical BoNT-A injection, which increased bladder capacity and decreased urgency sensation in patients with neurogenic or idiopathic detrusor overactivity (NDO, IDO). Excellent results were achieved with injection of either 100 U or 200 U of BoNT-A. Episodes of frequency, urgency, and UUI were reduced, maximal cystometric capacity increased, maximal detrusor pressure (Pdet) decreased, and the quality of life index also improved significantly. However, post void residual (PVR) volume increased significantly and some patients required clean intermittent catheterization (CIC) to evacuate the PVR. Dose-related adverse events (AE) increased with increasing dose of BoNT-A. Therefore, adjustments of the BoNT-A dose and sites of injection might minimize the de novo AE and help to maintain success rates.

DETAILED DESCRIPTION:
This study was designed as a single blind, randomized, parallel, actively controlled trial. The urodynamic DO confirmed patients were randomly assigned to receive injection of onabotulinumtoxinA 100 U (BoNT-A, Allergan, Irvine, California, USA), which was reconstituted to 10 ml with normal saline for suburothelial injections, in one of the three groups with the following injection number: (A) 100 U in 10ml injections, 1.0ml for each injection, totally 10 injections at bladder body (B) 100 U in 10ml, 0.5ml for each injection, totally 20 injections at bladder body, (C) 100 U in 10ml, 0.25ml for each injection, totally 40 injections at bladder body. Permuted block randomization was used for this trial. All treatments were evaluated at baseline and the primary end-point at 3 months.

The inclusion criteria were patients of either gender, aged 20 years or more, with urodynamic DO and at least one episode of urgency (urgency severity scale, USS≥2) or UUI per day as recorded in the 3-day voiding diary. Patients with neurogenic bladder, urodynamically confirmed bladder outlet obstruction, prior pelvic surgery, anti-incontinence surgery or urinary tract infection (UTI, white blood cell(WBC)>10/high power field (HPF) in urinalysis) were excluded. Informed consent was obtained from all patients before randomization. This study should be approved by the Institution Review Board and Ethics Committee of the hospital.

All patients had been managed with behavioral modification and treated with a certain number of antimuscarinics for more than 4 weeks before they were enrolled into this trial. Antimuscarinics was discontinued on the day of screening to wash out the remaining effect and obtaining a voiding diary that may reflect the true bladder condition.

The injection method for each patient was not recorded in the operation note and the study nurse who controlled the outcome measures was blinded to the treatment assignment. All procedures were performed transurethrally under intravenous general anesthesia in the operation room. Anticoagulant was discontinued 1 week prior to onabotulinumtoxinA treatment. The bladder volume was kept at 100-150 ml and the blood vessels were avoided during injections. An indwelling Foley catheter was placed in the bladder overnight and the patients were discharged the next morning. Broad-spectrum prophylactic antibiotics were given postoperatively for 3 days. Patients who developed acute urinary retention (AUR) or PVR volumes greater than 250 ml were advised to perform CIC periodically to evacuate their bladders. The patients were monitored at the outpatient clinic regularly for upto 24 months until symptoms returned to baseline levels.

Videourodynamic study was routinely performed at baseline, 3 and 6 months to measure urodynamic variables and detecting vesicoureteral reflux. The measured urodynamic variables included: maximum flow rate (Qmax), PVR, cystometric bladder capacity (CBC), detrusor pressure at Qmax (Pdet) and voiding efficiency (VE). The procedure and definition of videourodynamic study were in accordance of the recommendations of the International Continence Society.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients of either gender, aged 20 years or more, with urodynamic DO and at least one episode of urgency (urgency severity scale, USS≥2) or UUI per day as recorded in the 3-day voiding diary. Patients with neurogenic bladder, urodynamically confirmed bladder outlet obstruction, prior pelvic surgery, anti-incontinence surgery or urinary tract infection (UTI, white blood cell (WBC) >10/high power field (HPF) in urinalysis) were excluded. Informed consent was obtained from all patients before randomization. This study should be approved by the Institution Review Board and Ethics Committee of the hospital.

Exclusion Criteria:

* Use of antimuscarinic agent and effective in treatment of lower urinary tract symptoms
* Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up
* Patients with bladder outlet obstruction on enrollment
* Patients with postvoid residual > 150ml
* Patients with uncontrolled confirmed diagnosis of acute urinary tract infection
* Patients have laboratory abnormalities at screening including:
* Alanine aminotransferase (ALT)> 3 x upper limit of normal range
* Aspartate aminotransferase (AST)> 3 x upper limit of normal range
* Patients have abnormal serum creatinine level > 2 x upper limit of normal range
* Patients with any contraindication to be urethral catheterization during treatment
* Female patients who is pregnant, lactating, or with child-bearing potential without contraception.
* Myasthenia gravis, Eaton Lambert syndrome.
* Patients with any other serious disease considered by the investigator not suitable for general anesthesia or in the condition to enter the trial Patients participated investigational drug trial within 1 month before entering this study

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Global response assessment (GRA) of satisfaction by the patient | 2 weeks after initial treatment
  GRA (-3, -2, -1, 0, +1, +2, +3) of satisfaction by the patient
  * GRA≥+1: Respond
  * GRA≤0: Non-respond

SECONDARY OUTCOMES:
Voiding and urodynamic parameters | 2 weeks after the initial treatment day
  * Overactive bladder symptom score (OABSS)
  * Urgency severity score (USS)
  * Urgency urinary incontinence (UUI)/3 days
  * Urodynamic parameters
  * Functional bladder capacity (FBC)
  * Maximum flow rate (Qmax)
  * Postvoid residual volume (PVR)

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital and Tzu Chi University
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

REFERENCES:
- [Background] Abrams P, Kelleher CJ, Kerr LA, Rogers RG. Overactive bladder significantly affects quality of life. Am J Manag Care. 2000 Jul;6(11 Suppl):S580-90. PMID 11183901
- [Background] Irwin DE, Milsom I, Kopp Z, Abrams P, Cardozo L. Impact of overactive bladder symptoms on employment, social interactions and emotional well-being in six European countries. BJU Int. 2006 Jan;97(1):96-100. doi: 10.1111/j.1464-410X.2005.05889.x. PMID 16336336
- [Background] Milsom I, Abrams P, Cardozo L, Roberts RG, Thuroff J, Wein AJ. How widespread are the symptoms of an overactive bladder and how are they managed? A population-based prevalence study. BJU Int. 2001 Jun;87(9):760-6. doi: 10.1046/j.1464-410x.2001.02228.x. PMID 11412210
- [Background] Chen GD, Lin TL, Hu SW, Chen YC, Lin LY. Prevalence and correlation of urinary incontinence and overactive bladder in Taiwanese women. Neurourol Urodyn. 2003;22(2):109-17. doi: 10.1002/nau.10010. PMID 12579627
- [Background] Homma Y, Yamaguchi O, Hayashi K; Neurogenic Bladder Society Committee. An epidemiological survey of overactive bladder symptoms in Japan. BJU Int. 2005 Dec;96(9):1314-8. doi: 10.1111/j.1464-410X.2005.05835.x. PMID 16287452
- [Background] Kullmann FA, Artim DE, Birder LA, de Groat WC. Activation of muscarinic receptors in rat bladder sensory pathways alters reflex bladder activity. J Neurosci. 2008 Feb 20;28(8):1977-87. doi: 10.1523/JNEUROSCI.4694-07.2008. PMID 18287514
- [Background] Mukerji G, Yiangou Y, Grogono J, Underwood J, Agarwal SK, Khullar V, Anand P. Localization of M2 and M3 muscarinic receptors in human bladder disorders and their clinical correlations. J Urol. 2006 Jul;176(1):367-73. doi: 10.1016/S0022-5347(06)00563-5. PMID 16753445
- [Background] Ouslander JG. Management of overactive bladder. N Engl J Med. 2004 Feb 19;350(8):786-99. doi: 10.1056/NEJMra032662. No abstract available. PMID 14973214
- [Background] Dumoulin C, Hay-Smith J. Pelvic floor muscle training versus no treatment for urinary incontinence in women. A Cochrane systematic review. Eur J Phys Rehabil Med. 2008 Mar;44(1):47-63. PMID 18385628
- [Background] Simpson LL. Kinetic studies on the interaction between botulinum toxin type A and the cholinergic neuromuscular junction. J Pharmacol Exp Ther. 1980 Jan;212(1):16-21. PMID 6243359
- [Background] Apostolidis A, Popat R, Yiangou Y, Cockayne D, Ford AP, Davis JB, Dasgupta P, Fowler CJ, Anand P. Decreased sensory receptors P2X3 and TRPV1 in suburothelial nerve fibers following intradetrusor injections of botulinum toxin for human detrusor overactivity. J Urol. 2005 Sep;174(3):977-82; discussion 982-3. doi: 10.1097/01.ju.0000169481.42259.54. PMID 16094018
- [Background] Aoki KR. Evidence for antinociceptive activity of botulinum toxin type A in pain management. Headache. 2003 Jul-Aug;43 Suppl 1:S9-15. doi: 10.1046/j.1526-4610.43.7s.3.x. PMID 12887389
- [Background] Yiangou Y, Facer P, Ford A, Brady C, Wiseman O, Fowler CJ, Anand P. Capsaicin receptor VR1 and ATP-gated ion channel P2X3 in human urinary bladder. BJU Int. 2001 Jun;87(9):774-9. doi: 10.1046/j.1464-410x.2001.02190.x. PMID 11412212
- [Background] Avelino A, Cruz F. TRPV1 (vanilloid receptor) in the urinary tract: expression, function and clinical applications. Naunyn Schmiedebergs Arch Pharmacol. 2006 Jul;373(4):287-99. doi: 10.1007/s00210-006-0073-2. Epub 2006 May 24. PMID 16721555
- [Background] Popat R, Apostolidis A, Kalsi V, Gonzales G, Fowler CJ, Dasgupta P. A comparison between the response of patients with idiopathic detrusor overactivity and neurogenic detrusor overactivity to the first intradetrusor injection of botulinum-A toxin. J Urol. 2005 Sep;174(3):984-9. doi: 10.1097/01.ju.0000169480.43557.31. PMID 16094019
- [Background] Kuo HC. Urodynamic evidence of effectiveness of botulinum A toxin injection in treatment of detrusor overactivity refractory to anticholinergic agents. Urology. 2004 May;63(5):868-72. doi: 10.1016/j.urology.2003.12.007. PMID 15134967
- [Background] Sahai A, Khan MS, Dasgupta P. Efficacy of botulinum toxin-A for treating idiopathic detrusor overactivity: results from a single center, randomized, double-blind, placebo controlled trial. J Urol. 2007 Jun;177(6):2231-6. doi: 10.1016/j.juro.2007.01.130. PMID 17509328
- [Background] Brubaker L, Richter HE, Visco A, Mahajan S, Nygaard I, Braun TM, Barber MD, Menefee S, Schaffer J, Weber AM, Wei J; Pelvic Floor Disorders Network. Refractory idiopathic urge urinary incontinence and botulinum A injection. J Urol. 2008 Jul;180(1):217-22. doi: 10.1016/j.juro.2008.03.028. Epub 2008 May 21. PMID 18499184
- [Background] Reitz A, Stohrer M, Kramer G, Del Popolo G, Chartier-Kastler E, Pannek J, Burgdorfer H, Gocking K, Madersbacher H, Schumacher S, Richter R, von Tobel J, Schurch B. European experience of 200 cases treated with botulinum-A toxin injections into the detrusor muscle for urinary incontinence due to neurogenic detrusor overactivity. Eur Urol. 2004 Apr;45(4):510-5. doi: 10.1016/j.eururo.2003.12.004. PMID 15041117
- [Background] Kessler TM, Danuser H, Schumacher M, Studer UE, Burkhard FC. Botulinum A toxin injections into the detrusor: an effective treatment in idiopathic and neurogenic detrusor overactivity? Neurourol Urodyn. 2005;24(3):231-6. doi: 10.1002/nau.20105. PMID 15747344
- [Background] Rajkumar GN, Small DR, Mustafa AW, Conn G. A prospective study to evaluate the safety, tolerability, efficacy and durability of response of intravesical injection of botulinum toxin type A into detrusor muscle in patients with refractory idiopathic detrusor overactivity. BJU Int. 2005 Oct;96(6):848-52. doi: 10.1111/j.1464-410X.2005.05725.x. PMID 16153215
- [Background] Schulte-Baukloh H, Weiss C, Stolze T, Sturzebecher B, Knispel HH. Botulinum-A toxin for treatment of overactive bladder without detrusor overactivity: urodynamic outcome and patient satisfaction. Urology. 2005 Jul;66(1):82-7. doi: 10.1016/j.urology.2005.01.036. PMID 15992872
- [Background] Kuo HC. Clinical effects of suburothelial injection of botulinum A toxin on patients with nonneurogenic detrusor overactivity refractory to anticholinergics. Urology. 2005 Jul;66(1):94-8. doi: 10.1016/j.urology.2005.02.002. PMID 15992869
- [Background] Ghei M, Maraj BH, Miller R, Nathan S, O'Sullivan C, Fowler CJ, Shah PJ, Malone-Lee J. Effects of botulinum toxin B on refractory detrusor overactivity: a randomized, double-blind, placebo controlled, crossover trial. J Urol. 2005 Nov;174(5):1873-7; discussion 1877. doi: 10.1097/01.ju.0000177477.83991.88. PMID 16217327
- [Background] Sahai A, Sangster P, Kalsi V, Khan MS, Fowler CJ, Dasgupta P. Assessment of urodynamic and detrusor contractility variables in patients with overactive bladder syndrome treated with botulinum toxin-A: is incomplete bladder emptying predictable? BJU Int. 2009 Mar;103(5):630-4. doi: 10.1111/j.1464-410X.2008.08076.x. Epub 2008 Oct 16. PMID 18990156
- [Background] White WM, Pickens RB, Doggweiler R, Klein FA. Short-term efficacy of botulinum toxin a for refractory overactive bladder in the elderly population. J Urol. 2008 Dec;180(6):2522-6. doi: 10.1016/j.juro.2008.08.030. Epub 2008 Oct 19. PMID 18930481
- [Background] Brady CM, Apostolidis AN, Harper M, Yiangou Y, Beckett A, Jacques TS, Freeman A, Scaravilli F, Fowler CJ, Anand P. Parallel changes in bladder suburothelial vanilloid receptor TRPV1 and pan-neuronal marker PGP9.5 immunoreactivity in patients with neurogenic detrusor overactivity after intravesical resiniferatoxin treatment. BJU Int. 2004 Apr;93(6):770-6. doi: 10.1111/j.1464-410X.2003.04722.x. PMID 15049988
- [Background] Brady CM, Apostolidis A, Yiangou Y, Baecker PA, Ford AP, Freeman A, Jacques TS, Fowler CJ, Anand P. P2X3-immunoreactive nerve fibres in neurogenic detrusor overactivity and the effect of intravesical resiniferatoxin. Eur Urol. 2004 Aug;46(2):247-53. doi: 10.1016/j.eururo.2003.12.017. PMID 15245821
- [Background] Smet PJ, Moore KH, Jonavicius J. Distribution and colocalization of calcitonin gene-related peptide, tachykinins, and vasoactive intestinal peptide in normal and idiopathic unstable human urinary bladder. Lab Invest. 1997 Jul;77(1):37-49. PMID 9251677
- [Background] Yoshida M, Miyamae K, Iwashita H, Otani M, Inadome A. Management of detrusor dysfunction in the elderly: changes in acetylcholine and adenosine triphosphate release during aging. Urology. 2004 Mar;63(3 Suppl 1):17-23. doi: 10.1016/j.urology.2003.11.003. PMID 15013648
- [Background] Apostolidis A, Brady CM, Yiangou Y, Davis J, Fowler CJ, Anand P. Capsaicin receptor TRPV1 in urothelium of neurogenic human bladders and effect of intravesical resiniferatoxin. Urology. 2005 Feb;65(2):400-5. doi: 10.1016/j.urology.2004.10.007. PMID 15708075
- [Background] Wiseman OJ, Fowler CJ, Landon DN. The role of the human bladder lamina propria myofibroblast. BJU Int. 2003 Jan;91(1):89-93. doi: 10.1046/j.1464-410x.2003.03802.x. PMID 12614258
- [Background] Sui GP, Rothery S, Dupont E, Fry CH, Severs NJ. Gap junctions and connexin expression in human suburothelial interstitial cells. BJU Int. 2002 Jul;90(1):118-29. doi: 10.1046/j.1464-410x.2002.02834.x. PMID 12081783
- [Background] Apostolidis A, Dasgupta P, Fowler CJ. Proposed mechanism for the efficacy of injected botulinum toxin in the treatment of human detrusor overactivity. Eur Urol. 2006 Apr;49(4):644-50. doi: 10.1016/j.eururo.2005.12.010. Epub 2006 Jan 4. PMID 16426734
- [Background] Tyagi P, Wu PC, Chancellor M, Yoshimura N, Huang L. Recent advances in intravesical drug/gene delivery. Mol Pharm. 2006 Jul-Aug;3(4):369-79. doi: 10.1021/mp060001j. PMID 16889430
- [Background] Giannantoni A, Di Stasi SM, Chancellor MB, Costantini E, Porena M. New frontiers in intravesical therapies and drug delivery. Eur Urol. 2006 Dec;50(6):1183-93; discussion 1193. doi: 10.1016/j.eururo.2006.08.025. Epub 2006 Aug 30. PMID 16963179
- [Background] Giannantoni A, Porena M, Costantini E, Zucchi A, Mearini L, Mearini E. Botulinum A toxin intravesical injection in patients with painful bladder syndrome: 1-year followup. J Urol. 2008 Mar;179(3):1031-4. doi: 10.1016/j.juro.2007.10.032. Epub 2008 Jan 18. PMID 18206941
- [Background] Kuo HC, Liu HT, Yang WC. Therapeutic effect of multiple resiniferatoxin intravesical instillations in patients with refractory detrusor overactivity: a randomized, double-blind, placebo controlled study. J Urol. 2006 Aug;176(2):641-5. doi: 10.1016/j.juro.2006.03.087. PMID 16813911
- [Background] Birder LA. More than just a barrier: urothelium as a drug target for urinary bladder pain. Am J Physiol Renal Physiol. 2005 Sep;289(3):F489-95. doi: 10.1152/ajprenal.00467.2004. PMID 16093424
- [Background] Chuang YC, Yoshimura N, Huang CC, Chiang PH, Chancellor MB. Intravesical botulinum toxin a administration produces analgesia against acetic acid induced bladder pain responses in rats. J Urol. 2004 Oct;172(4 Pt 1):1529-32. doi: 10.1097/01.ju.0000137844.77524.97. PMID 15371885
- [Background] Liu HT, Chancellor MB, Kuo HC. Urinary nerve growth factor levels are elevated in patients with detrusor overactivity and decreased in responders to detrusor botulinum toxin-A injection. Eur Urol. 2009 Oct;56(4):700-6. doi: 10.1016/j.eururo.2008.04.037. Epub 2008 Apr 30. PMID 18472208
- [Background] Atiemo H, Wynes J, Chuo J, Nipkow L, Sklar GN, Chai TC. Effect of botulinum toxin on detrusor overactivity induced by intravesical adenosine triphosphate and capsaicin in a rat model. Urology. 2005 Mar;65(3):622-6. doi: 10.1016/j.urology.2004.10.057. PMID 15780404
- [Background] Crowley SL, Worchel FF, Ash MJ. Self-report, peer-report, and teacher-report measures of childhood depression: an analysis by item. J Pers Assess. 1992 Aug;59(1):189-203. doi: 10.1207/s15327752jpa5901_16. PMID 1512677
- [Background] Vemulakonda VM, Somogyi GT, Kiss S, Salas NA, Boone TB, Smith CP. Inhibitory effect of intravesically applied botulinum toxin A in chronic bladder inflammation. J Urol. 2005 Feb;173(2):621-4. doi: 10.1097/01.ju.0000143189.19835.f3. PMID 15643276
- [Background] Fraser MO, Chuang YC, Tyagi P, Yokoyama T, Yoshimura N, Huang L, De Groat WC, Chancellor MB. Intravesical liposome administration--a novel treatment for hyperactive bladder in the rat. Urology. 2003 Mar;61(3):656-63. doi: 10.1016/s0090-4295(02)02281-1. PMID 12639679
- [Background] Chuang YC, Tyagi P, Huang CC, Yoshimura N, Wu M, Kaufman J, Chancellor MB. Urodynamic and immunohistochemical evaluation of intravesical botulinum toxin A delivery using liposomes. J Urol. 2009 Aug;182(2):786-92. doi: 10.1016/j.juro.2009.03.083. Epub 2009 Jun 18. PMID 19539320
- [Background] Reimer K, Fleischer W, Brogmann B, Schreier H, Burkhard P, Lanzendorfer A, Gumbel H, Hoekstra H, Behrens-Baumann W. Povidone-iodine liposomes--an overview. Dermatology. 1997;195 Suppl 2:93-9. doi: 10.1159/000246039. PMID 9403264
- [Background] Egerdie RB, Reid G, Trachtenberg J. The effect of liposome encapsulated antineoplastic agents on transitional cell carcinoma in tissue culture. J Urol. 1989 Aug;142(2 Pt 1):390-8. doi: 10.1016/s0022-5347(17)38771-2. PMID 2501520
- [Background] Tyagi P, Chancellor MB, Li Z, De Groat WC, Yoshimura N, Fraser MO, Huang L. Urodynamic and immunohistochemical evaluation of intravesical capsaicin delivery using thermosensitive hydrogel and liposomes. J Urol. 2004 Jan;171(1):483-9. doi: 10.1097/01.ju.0000102360.11785.d7. PMID 14665960
- [Background] Chuang YC, Lee WC, Lee WC, Chiang PH. Intravesical liposome versus oral pentosan polysulfate for interstitial cystitis/painful bladder syndrome. J Urol. 2009 Oct;182(4):1393-400. doi: 10.1016/j.juro.2009.06.024. Epub 2009 Aug 15. PMID 19683290
- [Background] Liu HT, Kuo HC. Intravesical botulinum toxin A injections plus hydrodistension can reduce nerve growth factor production and control bladder pain in interstitial cystitis. Urology. 2007 Sep;70(3):463-8. doi: 10.1016/j.urology.2007.04.038. PMID 17905097
- [Background] Truschel ST, Wang E, Ruiz WG, Leung SM, Rojas R, Lavelle J, Zeidel M, Stoffer D, Apodaca G. Stretch-regulated exocytosis/endocytosis in bladder umbrella cells. Mol Biol Cell. 2002 Mar;13(3):830-46. doi: 10.1091/mbc.01-09-0435. PMID 11907265
- [Background] Wang E, Truschel S, Apodaca G. Analysis of hydrostatic pressure-induced changes in umbrella cell surface area. Methods. 2003 Jul;30(3):207-17. doi: 10.1016/s1046-2023(03)00027-6. PMID 12798135
- [Background] Cui M, Aoki KR. Botulinum toxin type A (BTX-A) reduces inflammatory pain in the rat formalin model. Cephalalgia 20:414-8, 2000.
- [Derived] Hsiao SM, Lin HH, Kuo HC. Factors Associated with Therapeutic Efficacy of Intravesical OnabotulinumtoxinA Injection for Overactive Bladder Syndrome. PLoS One. 2016 Jan 29;11(1):e0147137. doi: 10.1371/journal.pone.0147137. eCollection 2016. PMID 26824901